CLINICAL TRIAL: NCT04010669
Title: The Effect of Somatostatin in the Regulation of Velocity and Blood Flow of the Hepatic Circulation in Patients Undergoing Liver Resection
Brief Title: The Role of Somatostatin in the Hemodynamics of the Hepatic Circulation in Patients Undergoing Liver Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Kotsifa Evgenia, Principal Investigator, Laikο General Hospital, Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Somatostatin trial
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Portal Hypertension
Keywords: Portal Hypertension; Liver resection; Somatostatin
MeSH Terms: conditions — Hypertension, Portal | interventions — Somatostatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The study group includes participants who will receive somatostatin postoperatively (after liver resection).
  Interventions: Drug: Somatostatin
- Control group (Placebo Comparator): The control group includes participants who will receive placebo (a 24 hours infusion of 1000ml Normal Saline solution 0.9%) postoperatively (after liver resection).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatostatin — 2 amp of somatostatin at 1000ml normal saline solution in continuous 24-hour infusion for 5 days
  Arms: Study group
Drug: Placebo — 24 hours infusion of 1000ml Normal Saline solution 0.9%
  Arms: Control group

SUMMARY:
The purpose of the present clinical trial is to study the effect of somatostatin in the regulation of velocity and blood flow of the hepatic circulation in patients undergoing liver resection. The patients will be randomized in two groups: the study group will receive somatostatin and the control group will receive the placebo. In both groups, patients will undergo hepatectomy and directly postoperatively they will receive either somatostatin or placebo, depending on their randomization. The primary endpoint will be the increase or decrease of the velocity and the flow of the hepatic circulation estimated by ultrasonography compared to the same parameters when measured preoperatively.

DETAILED DESCRIPTION:
The purpose of the present clinical trial is to study the effect of somatostatin in the regulation of blood flow of the portal circulation at patients who have undergone hepatectomy. The patients will be randomized in two groups, namely the group that will receive somatostatin (study group) and the group that will receive the placebo (control group). In both groups, patients will undergo liver resection and directly postoperatively they will receive either somatostatin (2 amps at 1000ml normal saline solution in continuous 24-hour infusion for 5 days) or a 24 hours infusion of 1000ml Normal Saline solution 0.9%. On the first, third, fifth and seventh postoperative day, the velocity and the diameter of the portal vein, splenic vein, hepatic artery and hepatic veins will be measured sonographically and the flow will be calculated using the following mathematic formula: Flow= velocity x cross section area (the cross section area of the vessel can be calculated using the following equation: cross section area=πr2, with 'r' representing the vessel's radius).

Preoperatively

On the day before the surgery (day -1),an ultrasound will be performed in order to measure the velocity and the diameter of the portal vein, splenic vein, hepatic artery and hepatic veins and the flow will be calculated using the following mathematic formula: Flow= velocity x cross section area, as stated above. The following data will also be recorded: platelets, bilirubin (total and direct), albumin, cholesterol, urea, International Normalized Ratio, sodium, Serum Glutamic Oxaloacetic Transaminase, Serum Glutamic Pyruvic Transaminase, Alkaline Phosphatase, gamma-Glutamyl Transferase and the Model for End-stage Liver Disease score of each patient will be calculated. Finally, our patients will undergo a Computer Tomography scan in order to measure their liver and spleen volumetry.

On the day of the surgery

On the day of the surgery (day 0), the following information will be recorded: the type of the surgical procedure, the duration (in minutes), the presence of ascites, the number of times and total duration of the a pringle maneuver and finally the percentage of the resection of the parenchyma will be calculated. A biopsy of healthy liver tissue will be sent for histological examination in order to determine the presence of fibrosis/cirrhosis and its stage.

Postoperatively

On the first, third and fifth postoperative day (day 1, 3, 5), the preoperative blood test and the ultrasound measurements will be repeated and the amount of fluid in the drain(s) and inside the abdomen (via ultrasound) will be recorded. Finally, the fluid will be sent for biochemical examination and culture.

On the seventh postoperative day (day 7) all blood, fluid and ultrasound measurements will be repeated and also the liver and spleen volumetry via CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatectomy for any reason including primary malignant liver tumors (hepatocellular carcinomas, cholangiocellular carcinomas, etc), metastatic liver disease and symptomatic benign liver lesions (liver adenomas, focal nodular hyperplasia, hemangiomas, etc).
* Adult patients (≥18 years old)
* Patients whose indication for hepatectomy will be decided by a multidisciplinary team meeting.
* Patients who eill agree to sign an informed consent

Exclusion Criteria:

* Patients who do not meet the inclusion criteria and those
* Patients undergoing synchronous hepatectomy-colectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
The effect of somatostatin in the regulation of velocity of the hepatic circulation at patients who have undergone hepatectomy. | 7 days
  The velocity of the portal vein, splenic vein, hepatic artery and hepatic veins will be measured sonographically
The effect of somatostatin in the regulation of diameter of the vessels of the hepatic circulation at patients who have undergone hepatectomy. | 7 days
  The diameter of the portal vein, splenic vein, hepatic artery and hepatic veins will be measured sonographically
The effect of somatostatin in the regulation of blood flow of the hepatic circulation at patients who have undergone hepatectomy. | 7 days
  The blood flow of the portal vein, splenic vein, hepatic artery and hepatic veins will be calculated using the following mathematic formula: Flow= velocity x cross section area (the cross section area of the vessel can be calculated using the following equation: CSA=πr2, with 'r' representing the vessel's radius).

CONTACTS AND LOCATIONS:
Overall Officials: Georgios C Sotiropoulos, MD, PhD, Study Chair — Assistant Professor of Surgery, Laiko Hospital